CLINICAL TRIAL: NCT06883643
Title: Adoption of Innovative Approaches to Ensure Continuity of Quality TB Services During COVID-19 Pandemic in Lusaka and Livingstone, Zambia. (Telemedicine in TB)
Acronym: Telemed TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Ministry of Health, Zambia (Other Government); Centers for Disease Control and Prevention's COVID-19 Response International Task Force - CARES funding (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Telemedicine in TB; NU2GGH002251 (Other Grant/Funding Number: U.S. Centers for Disease Control and Prevention's COVID-19 Response International Task Force)
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Focus of the Study is to Evaluate DSD Models for Both TB Treatment and TPT Usiing Key Performance Indicators
Keywords: DSD TB

STUDY DESIGN:
Intervention Model Description: Project evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TB treatment ARM (Active Comparator): Beginning February 2022, we offered ATT via 2-month MMD during intensive and 4-month MMD during continuation phases.
  In-clinic visits during 6-months of ATT were reduced from 7 under standard of care to 3 visits in DSD, while ensuring robust adherence and adverse event screening.
  Remote monitoring consisted of structured SMS (months 1 to 5) and phone (week 2 and month 3) follow-up to assess adherence and screen for side effects. If SMS were not returned, a phone or home visit was triggered.
  Interventions: Behavioral: Differentiated service delivery approach (DSD) in TB treatment and prevention.
- TPT DSD (Active Comparator): Beginning February 2022, we offered TPT aligned to 6MMD ART model following standard of care processes with added support (See below).
  Remote monitoring consisted of structured SMS (months 1 to 5) and phone (week 2 and month 3) follow-up to assess adherence and screen for side effects.
  ROCs that did not respond to the SMS within 2 days were further contacted via phone and if not reachable a home visit was done.
  ROCs that reported at least one side effect or more were followed up with virtual reviews by clinicians.
  At enrollment ROCs reading language of preference was documented and the SMS was sent in their preferred language.
  Interventions: Behavioral: Differentiated service delivery approach (DSD) in TB treatment and prevention.

INTERVENTIONS:
Behavioral: Differentiated service delivery approach (DSD) in TB treatment and prevention. — Although DSD models have been widely adopted in HIV programs, DSD is a relatively new approach for TB programs because of an historical reliance on directly observed therapy (DOT) (6). DSD provides opportunities to improve health outcomes and reduce the burden of seeking care for people diagnosed with TB.

SUMMARY:
Following the negative impact of public health program services including TB services by the COVID-19 Pandemic in 2020, CIDRZ conducted a program evaluation for remote patient follow up for TB treatment and prevention through a differentiated service delivery model (DSD), offering clinical monitoring and psychosocial support while minimizing contact with the health facilities. The project was implemented between February 2022 to March 2023 and was funded through Centers for Disease Control and Prevention's COVID-19 Response International Task Force - CARES funding. While DSD models have been widely adopted in HIV programs , DSD is a relatively new and exciting approach for TB treatment and prevention programs.

DETAILED DESCRIPTION:
During the COVID-19 pandemic, government restrictions on movement decreased access to health care. Although DSD models have been widely adopted in HIV programs, this is a relatively new approach for TB programs. Zambia's NTLP has already changed policy to allow for such adaptations of service delivery, but these adaptations are not universally implemented and have not been evaluated at this time. This project aims to evaluate these DSD models for both TB treatment (Anti-TB Treatment ATT) and TPT using standardized indicators. To complement these DSD models, innovative approaches like digital (texting/SMS and phone) treatment support and remote monitoring of adverse events will be adopted using bi-directional SMS through use of the rapid pro system, a tool that allows medical information to be gathered and shared via a cell phone.

1. To implement TPT in 6MMD and ATT DSD models at 5 sites in Lusaka and Livingstone districts
2. To assess acceptability of TPT in 6MMD and ATT DSD models at implementation sties
3. To assess trends in TPT coverage and completion rates from pre-implementation through implementation periods using aggregate program performance data
4. To assess trends in ATT completion rates from pre-implementation through implementation periods using aggregate program performance data
5. To inform the Ministry of Health on a systematic approach for digital follow up and screening for TB and TPT RoCs aligned to MMD models of care.

ELIGIBILITY:
Inclusion Criteria:

TB ARM

* All ROCs presenting to chest clinic for TB treatment between February 2022 and September 2022 were considered for inclusion if:

Diagnosed with TB (new cases or retreatment cases) 18 years and above Willing and able to provide consent Not pregnant or breastfeeding No MDR TB

TPT ARM

All ROCs presenting to the ART clinic between February 2022 and September 2022 were considered for inclusion if they were:

18 years or above virally supressed with no symptoms or diagnosis suggestive of TB on ART for more than 6 months on 6MMD Consented to participate in the project did not receive TPT in the last 3 years not pregnant or breastfeeding women not incarcerated

Exclusion Criteria:

ATT ARM

* RoCs those TB diagnosis is not confirmed
* RoCs who are less than 18 years old
* RoCs not able to provide consent for program evaluation participation
* RoCs with MDR TB

TPT ARM

* RoCs with symptoms suggestive of TB, diagnosed or confirmed with TB diagnosis

  * RoCs who received TPT in the last 3 years
  * RoCs who are less than 18 years old
  * RoCs not able to provide consent for program evaluation participation
  * Pregnant and breastfeeding women
  * Incarcerated persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3318 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
TB and TPT Outcomes | 12 months
  • The primary program evaluation outcomes of interest are the TPT and ATT completion rates in the prospective cohort, defined as the fraction of participants completing TPT or ATT among those who initiated TPT or ATT

CONTACTS AND LOCATIONS:
Overall Officials: Mwanza Wa Mwanza, MD, Study Director — Centre for Infectious Disease Research in Zambia
Locations (1):
- Lusaka and Livingstone districts, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Differentiated Service Delivery — https://www.differentiatedcare.org/